CLINICAL TRIAL: NCT04350762
Title: Nutritional Supplementation in the Elderly With Weight Loss
Acronym: Elderly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll due to Pandemic
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Chief / Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-001995
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenia
Keywords: Elderly; protein supplementation; unintentional weight loss
MeSH Terms: conditions — Sarcopenia | interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement + Fish Oil (Experimental): Participants will mix 5 scoops of powdered nutrition supplement with 8 oz of cold water (2x/day). The supplemental shake will be consumed on two separate occasions daily. Omega-3 fish oil supplement is in capsule form for intake once daily.
  The NutraWell nutrition powder and OmegaRich fish oil supplement will be provided by and distributed from DoWell Laboratories (Irvine, CA - USA).
  Interventions: Dietary Supplement: Protein shake + Fish Oil
- Control (No Intervention): No dietary supplements. Participants will continue current intake.

INTERVENTIONS:
Dietary Supplement: Protein shake + Fish Oil — 2 shakes of protein as well as 1 fish oil daily.
  Arms: Supplement + Fish Oil

SUMMARY:
Many elderly experience weight loss and weakness with normal aging. Although there is extensive literature regarding nutritional advice for the elderly, there are few well- designed studies evaluating the effect of oral nutrition supplements in patients with weight loss and aging. The aim of this study is to examine the effect of dietary prescription with or without nutrition supplementation that includes soy protein, whey protein and fish oil in elderly patients who have suffered unintentional weight loss.

DETAILED DESCRIPTION:
This is an 8-week, randomized, pilot study with elderly subjects (age 65 and older) with recent unintentional weight loss who will receive either two servings of supplement powder and fish oil or no dietary supplementation (N=10 for each group).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 65 and older
* Non-smokers
* Weight loss >3% body weight over 6-12 months
* BMI ≤ 25
* Living independently or in an assisted living facility

Exclusion Criteria:

* Medical conditions that would lead to weight loss

  * Active cancer undergoing treatment (chemotherapy, radiation therapy, or planned surgical intervention)
  * CKD stage IV-V (eGFR <30) based on medical records within the last 12 months
  * Presence of dysphagia or odynophagia
  * Actively taking blood thinner such as Warfarin
  * Known history of cirrhosis with presence of ascites
  * History of a surgical procedure for weight loss (e.g. gastroplasty, gastric bypass, gastrectomy or partial gastrectomy, lap-band)
  * Any abnormal lab findings outside of normal limits as determined by the investigator
* Dietary conditions

  * Diet restrictions including vegetarianism, veganism, soy-free diet,
  * Fish and/or fish oil allergy or intolerance
  * Milk allergy excluding lactose intolerance
  * Follows a kosher diet
* Medications

  * Use of appetite stimulants (including megestrol, dronabinol and cyproheptadine).
  * Does not include medications used for depression (e.g. mirtazapine, paxil) if patient has been on a stable dose of this medication for at least 3 months prior to the start of this study
  * If participant is already taking a fish oil supplement, he/she must be willing to either stop the supplement or take the supplement the investigators are using in the study depending on the randomization assignment
* Additional

  * Patient has implantable device such as a pacemaker or ICD
  * Unable to complete 6-minute walk test at baseline
  * Hospitalization within the last 30 days
  * Participation in a therapeutic research study within 30 days of baseline
  * Living in a skilled nursing facility or long-term care facility
  * Any other medical condition that principal investigator or co-investigators deem would preclude the patient from study participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Body Composition | 8 weeks
  To assess if body composition is altered with increased protein supplementation using bioelectrical impedance body composition analysis to provide weight in pounds.
Nutritional Status | 8 weeks
  To assess if increased protein supplementation and fish oil has impact on nutrition status using Mini Nutritional Assessment questionnaire (minimum value 0, maximum value 14), where higher scores correlate to better nutritional status and lower scores indicate malnutrition.
Functional Improvements | 8 weeks
  To determine if protein supplementation improves functional movement using hand grip strength test as well as 6-minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, 1000 Veteran Ave., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No